CLINICAL TRIAL: NCT04280159
Title: Modern Hybrid Imaging for Staging and Monitoring Patients With Oral Squamous Cell Carcinoma
Brief Title: Modern Hybrid Imaging in Patients With OSCC
Acronym: PETOSCC
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PETOSCC
Record Dates: First submitted 2020-02-04; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Neoplasm
Keywords: Head and Neck; SCC; PET/CT; Staging
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective diagnostic study to determine the diagnostic accuracy of preoperative 18F--fluorodeoxyglucose (FDG) positron emission tomography/computed tomography (PET/CT) in detecting local tumor extent, cervical lymph node metastases and distant metastases/secondary primary tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological proven head and neck carcinoma
* Written inform consent
* 18 years of age

Exclusion Criteria:

* Cancer of unknown primary
* En-bloc resection of lymph node levels
* Uncertainties regarding the removed lymph node levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with squamous cell carcinoma of the oral cavity,
Sampling Method: Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of FGD-PET/CT to detect the primary tumor | 2013-2018
  Visual assessment of FDG-PET/CT will be performed according to current guidelines. The localization, expansion, and infiltration of osseous structures will be recorded. The outcome measure is the correct diagnosis (1 = correct; 0 = false) with regards to the histopathological analysis. The outcome measure will then be used to calculate the diagnostic accuracy of FDG-PET/CT to detect the primary tumor.
Diagnostic accuracy of FGD-PET/CT to detect lymph nodes metastases | 2013-2018
  Visual assessment of FDG-PET/CT will be performed according to current guidelines. The presence and number of nodal metastasis will be recorded for each cervical lymph node level. The outcome measure is the correct diagnosis (1 = correct; 0 = false) with regards to the histopathological analysis. The analysis will be performed on a patient level (lymph node metastasis yes/no), on the nodal metastatic involvement of cervical sides and lymph node levels. The outcome measure will then be used to calculate the diagnostic accuracy of FDG-PET/CT to detect lymph node metastases.
Diagnostic accuracy of FGD-PET/CT to detect distant lymph node metastases. | 2013-2018
  Visual assessment of FDG-PET/CT will be performed according to current guidelines. The presence, localization and number of distant nodal metastasis will be recorded. The outcome measure is the correct diagnosis (1 = correct; 0 = false) with regards to the histopathological analysis. The outcome measure will then be used to calculate the diagnostic accuracy of FDG-PET/CT to detect lymph node metastases.

SECONDARY OUTCOMES:
Diagnostic accuracy of MRI to detect the primary tumor | 2013-2018
  Visual assessment of MRI will be performed according to current guidelines. The localization, expansion, and infiltration of osseous structures will be recorded. The outcome measure is the correct diagnosis (1 = correct; 0 = false) with regards to the histopathological analysis. The outcome measure will then be used to calculate the diagnostic accuracy of MRI to detect the primary tumor.
Diagnostic accuracy of MRI to detect lymph nodes metastases | 2013-2018
  Visual assessment of MRI will be performed according to current guidelines. The presence and number of nodal metastasis will be recorded for each cervical lymph node level. The outcome measure is the correct diagnosis (1 = correct; 0 = false) with regards to the histopathological analysis. The analysis will be performed on a patient level (lymph node metastasis yes/no), on the nodal metastatic involvement of cervical sides and lymph node levels. The outcome measure will then be used to calculate the diagnostic accuracy of MRI to detect lymph node metastases.
Diagnostic accuracy of CT to detect the primary tumor | 2013-2018
  Visual assessment of CT will be performed according to current guidelines. The localization, expansion, and infiltration of osseous structures will be recorded. The outcome measure is the correct diagnosis (1 = correct; 0 = false) with regards to the histopathological analysis. The outcome measure will then be used to calculate the diagnostic accuracy of CT to detect the primary tumor.
Diagnostic accuracy of CT to detect lymph nodes metastases | 2013-2018
  Visual assessment of CT will be performed according to current guidelines. The presence and number of nodal metastasis will be recorded for each cervical lymph node level. The outcome measure is the correct diagnosis (1 = correct; 0 = false) with regards to the histopathological analysis. The analysis will be performed on a patient level (lymph node metastasis yes/no), on the nodal metastatic involvement of cervical sides and lymph node levels. The outcome measure will then be used to calculate the diagnostic accuracy of CT to detect lymph node metastases.
Diagnostic accuracy of CT to detect distant lymph node metastases. | 2013-2018
  Visual assessment of CT will be performed according to current guidelines. The presence, localization and number of distant nodal metastasis will be recorded. The outcome measure is the correct diagnosis (1 = correct; 0 = false) with regards to the histopathological analysis. The outcome measure will then be used to calculate the diagnostic accuracy of CT to detect lymph node metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Urs Müller-Richter, MD, DDS, PhD, Principal Investigator — Dpt. of CMF, University Hospital Wuerzburg
Locations (1):
- Department of Cranio- and Maxillofacial Surgery, Würzburg, Germany